CLINICAL TRIAL: NCT01869504
Title: A Feasibility and Safety Study of the Use of a Dedicated Ballooned Intercostal Drain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sherwood Forest Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SFH1
Record Dates: First submitted 2013-02-26; First posted 2013-06-05 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Pleural Effusion
Keywords: Ballooned intercostal drain; Pleural effusion
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Balloon-tipped intercostal drain (Experimental): Subjects who have given written informed consent and who fulfill the inclusion and exclusion criteria will proceed to have the study drain inserted at the earliest opportunity as per standard hospital protocols using local anaesthetic, and conscious sedation where appropriate. All other aspects of their treatment will be identical to usual clinical care, including chest drain checks and fluid drainage strategies.
  Interventions: Device: Balloon-tipped intercostal drain

INTERVENTIONS:
Device: Balloon-tipped intercostal drain — Ballooned intercostal drain for pleural effusion, inserted using local anaesthetic and ultrasound guidance.
  Other Names: Manufactured by Rocket Medical.

SUMMARY:
Drainage of air and fluid from the chest cavity using plastic tubes (chest drains) is an essential tool in Chest Medicine. A common complication of drain insertion is accidental removal of the drain, usually as a result of inadequate securing techniques, with rates of up to 1 in 5 reported. This often results in the need for further procedures (including drain re-siting), with associated additional risk to the patient and an increase in health care costs. One suggested method to reduce premature drain removal is to use chest drains with ballooned tips, much like a bladder catheter. These would provide a physical obstruction inside the chest cavity at the insertion site, whilst being easy to use as stitching or extensive taping may not be required.

The investigators propose a trial of a dedicated ballooned chest drain to investigate whether a reduction in drain re-siting rates can be achieved. Pain scores will also be assessed during this trial to ensure that irritation of the lining of the lung or chest wall by the balloon is not excessive.

ELIGIBILITY:
Inclusion Criteria:

* Age >16 years
* Able to give written informed consent
* Requiring intercostal tube drainage of a pleural effusion for clinical reasons

Exclusion Criteria:

* Requiring intercostal tube drainage for chest trauma
* Requiring blunt dissection for drain insertion

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The percentage of intercostal drains requiring re-siting | 7 days
  It is likely that most if not all of the drains will have been removed by this time owing to resolution of the effusion, but the time period of 7 days has been selected to allow maximum data capture.

SECONDARY OUTCOMES:
Patient reported pain scores, using a visual analogue scale | At 24 hours, 72 hours, and at drain removal, an expected average of 5 days
The frequency of balloon rupture | 7 days
  It is likely that most if not all of the drains will have been removed by this time owing to resolution of the effusion, but the time period of 7 days has been selected to allow maximum data capture.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel V Kemp, MBBS, Principal Investigator — Sherwood Forest Hospitals NHS Foundation Trust
Locations (1):
- King's Mill Hospital, Sutton in Ashfield, Nottinghamshire, United Kingdom